CLINICAL TRIAL: NCT02937870
Title: A Proof of Principle Bite Force Study Using Two New Test Adhesives and a Currently Marketed Denture Adhesive.
Brief Title: A Bite Force Study Comparing Two New Test Adhesives With Currently Marketed Denture Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 206233
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-02

CONDITIONS: Denture Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Test Product 1 (Experimental): Applied topically to upper denture, to clean dry denture fit surface in a pattern consistent with application instructions.
  Interventions: Device: Test Product 1
- Test Product 2 (Experimental): Applied topically to upper denture, to clean dry denture fit surface in a pattern consistent with application instructions.
  Interventions: Device: Test Product 2
- Reference Product (Active Comparator): Applied topically to upper denture, to clean dry denture fit surface in a pattern consistent with application instructions.
  Interventions: Device: Reference Product
- Negative Control (Other)
  Interventions: Other: Negative Control

INTERVENTIONS:
Device: Test Product 1 — Test adhesive 1 with a thin nozzle
  Arms: Test Product 1
Device: Test Product 2 — Test adhesive 2 with a thin nozzle
  Arms: Test Product 2
Device: Reference Product — Adhesive Cream
  Arms: Reference Product
Other: Negative Control — No adhesive
  Arms: Negative Control

SUMMARY:
The objective of this 4-treatment, 4-period, randomized, crossover, proof of principle bite force study will be to compare bite force measurements over a 12 hour period across two (test) cream denture adhesives, with a currently marketed cream denture adhesive (positive control), and a negative/no treatment control.

DETAILED DESCRIPTION:
This will be a 4-treatment, 4-period, randomized, crossover, proof of principle bite force study which will compare bite force measurements over a 12 hour period across two cream denture adhesives with a currently marketed cream denture adhesive (positive control), and a negative/no treatment control. A short questionnaire regarding the flavor and texture characteristics of each denture adhesive after a single use will also be administered to give an indication of participant satisfaction of these attributes.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18 to 85 years.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities in medical history or upon oral examination and absence of any condition that could affect the participant's safety or wellbeing or their ability to understand and follow study procedures and requirements.
* Completely edentulous maxillary arch restored with a conventional full acrylic based upper complete denture. Dentate, partial or full edentulous mandibular arch. Partial or full edentulous arch may be restored with a stable complete, partial or implant supported denture. Maxillary dentures must be considered to be moderately well-fitting at the screening visit (Kapur Index, Olshan Modification: retention score >=2, stability score >=2). Maxillary dentures and mandibular dentures, if present, must be considered to be well-made based on design and construction criteria specified in the protocol. The qualifying maxillary incisal bite force readings (without adhesive) must be less than or equal to 9 pounds (lb) at the Screening Visit and subsequent visit pre-treatment baseline bites. At least 2 of the 4 qualifying bite readings at the Screening Visit must be reproducible (+/- 2lb). At subsequent visits the bite force readings must be within +/-2lb for 1 of the 3 practice bites and the pre-treatment baseline bite.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.

Exclusion Criteria:

* A woman who is known to be pregnant or who is intending to become pregnant (self reported) over the duration of the study.
* A woman who is breast-feeding.
* Implanted with a cardiac pacemaker.
* Daily doses of medication that might interfere with the ability to perform the study according to protocol (as determined by the Investigator).
* Taking or have taken a bisphosphonate drug for treatment of osteoporosis.
* A serious chronic disease requiring hospitalization.
* Any condition not previously mentioned that in the Investigator's opinion may impair the study evaluation.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Any clinically significant or relevant oral abnormality (e.g. temporomandibular joint [TMJ] problems) that, in the opinion of the investigator, could affect the participant's participation in the study.
* Any participant clinically identified as having an incisal bite relation which could affect the bite force measurements.
* Severe dry mouth that may affect denture retention in the opinion of the Investigator.
* OST examination findings such as stomatitis, open sores, lesions, redness or swelling that, in the opinion of the investigator, could affect the participant's participation in the study.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* A participant who is unwilling to refrain from smoking, including e-cigarettes and the use of chewing tobacco or other tobacco products for the duration of screening and each treatment day (12-14 hours).
* An employee of the sponsor or the study site or members of their immediate family.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bloomfield, New Jersey, United States

REFERENCES:
- [Derived] Atassi M, Ling MR, Oneglia K, Dilauro TS. A proof-of-principle bite force study using two experimental test denture adhesives and a currently marketed denture adhesive. Clin Exp Dent Res. 2020 Apr;6(2):266-273. doi: 10.1002/cre2.256. Epub 2020 Feb 6. PMID 32026625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single center in USA.
Pre-assignment Details: A total of 37 participants were screened. Out of which 23 participants were randomized in the study. 14 participants were not randomized in the study because 12 of which were screened failure, one participant withdrew consent and one participant was dismissed because number of participants required being reached.
Groups:
- Overall Study: This was a single-center, randomized, controlled, examiner-blind, four-treatment, four-period, crossover study. Participants received a single application of each study treatment, lasting for 12 hours.
Period: Overall Study
Arm/Group | Overall Study
Started | 23
Received Test Adhesive 1 | 21
Received Test Adhesive 2 | 22
Received Positive Control Adhesive | 21
Received no Adhesive | 20
Completed | 20
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Protocol Deviation | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Participants: All randomized participants who received all four treatments: test adhesive 1, test adhesive 2, positive control adhesive and no adhesive were included in the baseline assessment.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Over Baseline Over 12 Hours (AOB0-12) for Test Adhesive 1 Versus (vs.) No Adhesive
Description: Area over baseline over 12 hours (AOB0-12) was assessed to measure the incisal bite force. AOB0-12 was calculated as area under the curve over 12 hours [AUC0-12])/12 hours minus baseline bite force (pounds [lbs]). AUC0-12 was calculated using the trapezoidal method. This transformation returned the measurement to the same scale as the original observations. Higher values of AOB0-12 demonstrate a stronger bite force overtime than lower values.
Time Frame: up to 12 hours
Population: Analysis for this outcome was performed on intent-to-treat (ITT) population which included all randomized participants with at least one post baseline assessment of efficacy. Number of participants analyzed are the participants from ITT population analyzed for this outcome.
Measure: Least Squares Mean (Standard Error); unit: lbs
Groups:
- Test Adhesive 1: Participants of this arm topically applied test adhesive 1 to upper denture, to clean dry denture fit surface in a pattern consistent with application instructions.
- No Adhesive: Participants of this arm did not receive any adhesive to apply on upper denture.
Arm/Group | Test Adhesive 1 | No Adhesive
Number analyzed (Participants) | 20 | 20
lbs | 2.09 (0.34) | 1.43 (0.33)
Statistical Analysis 1: Comparison: Test Adhesive 1 vs No Adhesive; Test type: Other; p = 0.1770, ANCOVA — p-values for treatment comparison of test adhesive 1 vs. no adhesive were adjusted using the Dunnett's method; ANCOVA with factors for subject (random effect), period & treatment, subject-level and period-level pre-treatment baseline bite force as covariate; Least square (LS) mean difference = 0.66, 95% CI 2-sided [-0.14 to 1.47] — Difference is first-named treatment minus second-named treatment such that a positive difference favours the first named treatment

2. Primary Outcome: Area Over Baseline Over 12 Hours (AOB0-12) for Test Adhesive 2 vs. No Adhesive
Description: Area over baseline over 12 hours (AOB0-12) was assessed to measure the incisal bite force. AOB0-12 was calculated as area under the curve over 12 hours [AUC0-12])/12 hours minus baseline bite force (lbs). AUC0-12 was calculated using the trapezoidal method. This transformation returned the measurement to the same scale as the original observations. Higher values of AOB0-12 demonstrate a stronger bite force overtime than lower values.
Time Frame: up to 12 hours
Population: Analysis for this outcome was performed on ITT population which included all randomized participants with at least one post baseline assessment of efficacy. Number of participants analyzed are the participants from ITT population analyzed for this outcome.
Measure: Least Squares Mean (Standard Error); unit: lbs
Groups:
- Test Adhesive 2: Participants of this arm topically applied test adhesive 2 to upper denture, to clean dry denture fit surface in a pattern consistent with application instructions.
Arm/Group | Test Adhesive 2 | No Adhesive
Number analyzed (Participants) | 21 | 20
lbs | 1.23 (0.33) | 1.43 (0.33)
Statistical Analysis 1: Comparison: Test Adhesive 2 vs No Adhesive; Test type: Other; p = 0.8321, ANCOVA — p-values for treatment comparison of test adhesive 1 vs. no adhesive were adjusted using the Dunnett's method; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.20, 95% CI 2-sided [-0.98 to 0.59] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Over Baseline Over 12 Hours (AOB0-12) for Test Adhesive 1 vs. Positive Control Adhesive
Description: as for outcome 2
Time Frame: up to 12 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: lbs
Groups:
- Positive Control Adhesive: Participants of this arm topically applied commercial denture adhesive to upper denture, to clean dry denture fit surface in a pattern consistent with application instructions.
Arm/Group | Test Adhesive 1 | Positive Control Adhesive
Number analyzed (Participants) | 20 | 20
lbs | 2.09 (0.34) | 2.02 (0.33)
Statistical Analysis 1: Comparison: Test Adhesive 1 vs Positive Control Adhesive; Test type: Other; p = 0.8566, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.07, 95% CI 2-sided [-0.72 to 0.87] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Area Over Baseline Over 12 Hours (AOB0-12) for Test Adhesive 2 vs. Positive Control Adhesive
Description: as for outcome 2
Time Frame: up to 12 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: lbs
Groups:
- Test Adhesive 2: Participants of this arm received topical application of test adhesive 2 to upper denture by site study staff, to clean dry denture fit surface in a pattern consistent with application instructions.
- Positive Control Adhesive: Participants of this arm received topical application of commercial adhesive to upper denture by site study staff, to clean dry denture fit surface in a pattern consistent with application instructions.
Arm/Group | Test Adhesive 2 | Positive Control Adhesive
Number analyzed (Participants) | 21 | 20
lbs | 1.23 (0.33) | 2.02 (0.33)
Statistical Analysis 1: Comparison: Test Adhesive 2 vs Positive Control Adhesive; Test type: Other; p = 0.0488, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.79, 95% CI 2-sided [-1.58 to -0.00] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Area Over Baseline Over 12 Hours (AOB0-12) for Test Adhesive 1 vs. Test Adhesive 2
Description: as for outcome 2
Time Frame: up to 12 hours
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: lbs
Groups:
- Test Adhesive 1: Participants of this arm received topical application of test adhesive 1 to upper denture by site study staff, to clean dry denture fit surface in a pattern consistent with application instructions.
Arm/Group | Test Adhesive 1 | Test Adhesive 2
Number analyzed (Participants) | 20 | 21
lbs | 2.09 (0.34) | 1.23 (0.33)
Statistical Analysis 1: Comparison: Test Adhesive 1; Test type: Other; p = 0.0352, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference = 0.86, 95% CI 2-sided [0.06 to 1.66] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: up to 61 days (AEs were collected from OST examination from screening to last study visit)
Groups:
- Negative Control: Participants of this arm did not receive any adhesive to apply on upper denture.
Arm/Group | Test Adhesive 1 | Test Adhesive 2 | Positive Control Adhesive | Negative Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 1/21 | 3/22 | 2/21 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Adhesive 1 (N=21) | Test Adhesive 2 (N=22) | Positive Control Adhesive (N=21) | Negative Control (N=20)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT02937870/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT02937870/SAP_001.pdf